CLINICAL TRIAL: NCT01122693
Title: A Prospective, Randomized Comparison Between Two Ultrasound Technologies for Ultrasound-guided Catheter Placement in Regional Anesthesia
Brief Title: Comparison Between Two Ultrasound Technologies for Ultrasound-guided Catheter Placement in Regional Anesthesia
Acronym: eZono
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Univ. Prof. Dr. med. Claudia Spies, Department of Anesthesiology and Operative Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: eZono
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Anesthesia
Keywords: Regional Anesthesia; Pain Medicine; Ultrasound; Nerve Blocks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard 2D ultrasound images (Active Comparator)
  Interventions: Device: eZono - high-quality 2D ultrasound images; Device: standard 2D ultrasound images
- high-quality 2D ultrasound images (Experimental)
  Interventions: Device: eZono - high-quality 2D ultrasound images; Device: standard 2D ultrasound images
- nerve stimulation techniques (Active Comparator)
  Interventions: Device: eZono - high-quality 2D ultrasound images; Device: standard 2D ultrasound images

INTERVENTIONS:
Device: eZono - high-quality 2D ultrasound images — higher ultrasound frequencies, better image resolution, better post-processing and user-friendliness.
Device: standard 2D ultrasound images — current standard in two-dimensional (2D) ultrasound images

SUMMARY:
The use of ultrasound imaging techniques in regional anaesthesia is rapidly becoming an area of increasing interest. It represents one of the largest changes that the field of regional anaesthesia has seen. For the first time, the operator is able to view an image of the target nerve directly, guide the needle under real-time observation, navigate away from sensitive anatomy, and monitor the spread of local anaesthetic (LA).The key to successful regional anaesthesia is deposition of LA accurately around the nerve structures.

In the past, electrical stimulation which relied on surface landmark identification, was used for this. However, landmark techniques have limitations; variations in anatomy and nerve physiology , as well as equipment accuracy have had an effect on success rates and complications.

However, alongside the enthusiasm of ultrasound guidance in regional anaesthesia, there should be a degree of informed scepticism. The widespread use of the various techniques of ultrasound-guided regional blocks without adequate training raises the danger of malpractice and subsequent impaired outcome.

Adequate education in the use of regional block techniques under ultrasound guidance is essential. Recent technical developments have achieved higher ultrasound frequencies and better image resolution, as well as better post-processing and user-friendliness.

The purpose of this study is to determine whether new technical features such as reference images, higher ultrasound frequencies, better image resolution and smaller size and weight of the ultrasound probes may improve outcome (clinical benefits) and may show an increased efficacy and safety. And if the new technology of ultrasound images improves the training quality of trainees and novices in the art of ultrasound-guided blocks.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the age of 18 and above who need a regional anesthesia catheter for postoperative pain management after elective orthopedic surgery

Exclusion Criteria:

* Participation in another trial according to the German Drug Law 30 days to and during the study
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Absent knowledge of German language
* Analphabetism
* Allergy to local anesthesia or other ingredients of the intravenous solutions
* For women: Pregnancy or positive pregnancy test within the preoperative screening
* Operation due to case of emergency, polytrauma or pathologic fracture
* American Society of Anaesthesiologists (ASA) classification greater than III
* Peripheral or central edema
* AIDS (according to the CDC-classification of HIV-infection: category C)
* Immunosuppression therapy
* History of bleeding tendency (e.g. von-Willebrand-disease, thrombocytopenia)
* Derailed metabolic disorder (e.g. Diabetes mellitus (Glucose > 300 mg/dl) during the preoperative screening)
* Known history of electrolyte disturbance (e.g. Hyperkalemia > 5.8 mmol/l, Hypernatraemia > 155 mmol/l)
* Known history of acid-base-dysbalances
* History of intracranial hemorrhage within one year of participation in the study
* Neurological or psychiatric disease with limited contractual capability
* CHF (congestive heart failure) according to (New York Heart Association) classification - NYHA class IV
* Liver disease (CHILD B or C cirrhosis, end-stage liver disease (MELD-score greater than 10)
* Renal insufficiency (serum creatinine greater than 2.0 mg/dl or greater than 150 µmol/l or dependency of haemodialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Reduction in time to perform the catheter placement in regional anesthesia | first three days

SECONDARY OUTCOMES:
Improvement in performance: Incidence of complications | first three days
Improvement of success rate regarding correct catheter placement | first three days

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Klinik für Anästhesiologie, Berlin, State of Berlin
  - Department of Anesthesiology and Operative Intensive Care Medicine Campus Charité Mitte / Campus Virchow-Klinikum, Berlin, State of Berlin